CLINICAL TRIAL: NCT05540522
Title: A PHASE 3, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE EFFICACY, SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MODIFIED RNA VACCINE AGAINST INFLUENZA COMPARED TO LICENSED INACTIVATED INFLUENZA VACCINE IN HEALTHY ADULTS 18 YEARS OF AGE OR OLDER
Brief Title: A Study to Evaluate a Modified RNA Vaccine Against Influenza in Adults 18 Years of Age or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4781004; NCT05540522 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Influenza, Human
Keywords: Grippe; Flu; Influenza; Vaccine; RNA vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Quadrivalent influenza modRNA vaccine, 18 through 64 years of age (Experimental): Quadrivalent influenza modRNA vaccine (single dose), participants 18 through 64 years of age
  Interventions: Biological: Quadrivalent influenza modRNA vaccine
- Quadrivalent influenza vaccine, 18 through 64 years of age (Active Comparator): Licensed quadrivalent influenza vaccine (single dose), participants 18 through 64 years of age
  Interventions: Biological: Quadrivalent influenza vaccine
- Quadrivalent influenza modRNA vaccine, ≥65 years of age (Experimental): Quadrivalent influenza modRNA vaccine (single dose), participants ≥65 years of age
  Interventions: Biological: Quadrivalent influenza modRNA vaccine
- Quadrivalent influenza vaccine, ≥65 years of age (Active Comparator): Licensed quadrivalent influenza vaccine (single dose), participants ≥65 years of age
  Interventions: Biological: Quadrivalent influenza vaccine

INTERVENTIONS:
Biological: Quadrivalent influenza modRNA vaccine — Quadrivalent influenza modRNA vaccine (single dose)
  Arms: Quadrivalent influenza modRNA vaccine, 18 through 64 years of age; Quadrivalent influenza modRNA vaccine, ≥65 years of age
Biological: Quadrivalent influenza vaccine — Licensed quadrivalent influenza vaccine (single dose)
  Arms: Quadrivalent influenza vaccine, 18 through 64 years of age; Quadrivalent influenza vaccine, ≥65 years of age

SUMMARY:
This is a Phase 3, randomized, observer-blinded study to evaluate the efficacy, safety, tolerability, and immunogenicity of a single dose of a quadrivalent influenza modRNA vaccine compared to licensed inactivated influenza vaccine in healthy adults 18 years of age and older.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, observer-blinded study to evaluate the efficacy, safety, tolerability, and immunogenicity of a quadrivalent influenza modRNA vaccine (qIRV) encoding HA of 4 seasonally recommended strains (2 A strains and 2 B strains) compared to licensed quadrivalent influenza vaccine (QIV) in healthy adults 18 years of age and older.

Participants may be enrolled in either the reactogenicity subset, immunogenicity subset, or both/neither subset(s). Efficacy will be assessed in this study through surveillance for influenza-like illness.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years of age at Visit 1 (Day 1).
2. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
4. Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
3. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
4. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
5. Allergy to egg proteins (egg or egg products) or chicken proteins.
6. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), eg, for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
7. Receipt of blood/plasma products or immunoglobulin from 60 days before study intervention administration, or planned receipt throughout the study.
8. Vaccination with any investigational or licensed influenza vaccine within 6 months (175 days) before study intervention administration, or ongoing receipt of chronic antiviral therapy with activity against influenza.
9. Any participant who has received or plans to receive a modRNA-platform SARS CoV-2 vaccine within 14 days before or after study vaccination at Visit 1.
10. Participation in other studies involving administration of a study intervention within 28 days prior to, and/or during, participation in this study.
11. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45789 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (318):
- United States (260):
  - North Alabama Research Center, Athens, Alabama
  - St. Vincent's Birmingham Hospital, Birmingham, Alabama
  - Accel Research Sites Network - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Ross Bridge Medical Practice, LLC-CCT Research, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Lenzmeier Family Medicine/CCT Research, Glendale, Arizona
  - Aventiv Research, Mesa, Arizona
  - Desert Clinical Research/ CCT Research, Mesa, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - HOPE Research Institute - Phoenix, Phoenix, Arizona
  - Foothills Research Center/ CCT Research, Phoenix, Arizona
  - Epic Medical Research - Surprise, Surprise, Arizona
  - Fiel Family and Sports Medicine, PC/CCT Research, Tempe, Arizona
  - HOPE Research Institute, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Baptist Health Center For Clinical Research, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Velocity Clinical Research, San Bernardino, Banning, California
  - Benchmark Research, Colton, California
  - Ascada Health PC dba Ascada Research, Fullerton, California
  - Marvel Clinical Research, Huntington Beach, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Orange County Research Center, Lake Forest, California
  - Ark Clinical Research, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Empire Clinical Research, Pomona, California
  - Paradigm Clinical Research Centers, Inc, Redding, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Benchmark Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Wr-McCr, Llc, San Diego, California
  - California Research Foundation, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Ark Clinical Research - Tustin, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Tekton Research, LLC., Fort Collins, Colorado
  - Tekton Research, LLC., Longmont, Colorado
  - Paradigm Clinical Research Centers, Inc, Wheat Ridge, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Clinical Research Consulting, Milford, Connecticut
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Yale Cardiology, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Washington Health Institute, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Robert B. Pritt, DO, Fort Myers, Florida
  - Best Quality Research,Inc., Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Health Awareness, Jupiter, Florida
  - Wr-Msra.Llc, Lake City, Florida
  - JEM Research Institute, Lake Worth, Florida
  - Accel Research Sites Network - Lakeland Clinical Research Unit, Lakeland, Florida
  - Accel Research Sites - St. Petersburg Clinical Research Unit, Largo, Florida
  - Accel Research Sites Network - Maitland Clinical Research Unit, Maitland, Florida
  - Care Research - West Flagler Street, Miami, Florida
  - Gerardo Polanco, MD, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - United Medical Research, Port Orange, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - IACT Health, Rincon, Georgia
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - AGILE Clinical Research Trials, LLC, Sandy Springs, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Javara - Privia Medical Group Georgia - Savannah, Savannah, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Prime, Idaho Falls, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Koch Family Medicine, Morton, Illinois
  - Accellacare - DuPage, Oak Lawn, Illinois
  - MediSphere Medical Research Center - Evansville - West Franklin Street, Evansville, Indiana
  - MediSphere Medical Research Center - EAST, Evansville, Indiana
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - University of Iowa, Iowa City, Iowa
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Versailles Family Medicine / CCT Research, Versailles, Kentucky
  - MedPharmics, LLC, Lafayette, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Pharmaron, Baltimore, Maryland
  - Advanced Primary and Geriatric Care - CCT Research, Rockville, Maryland
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Grosse Pointe Woods, Michigan
  - Revival Research Institute, LLC, Sterling Heights, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Bio-Kinetic Clinical Applications, LLD dba QPS-MO, Springfield, Missouri
  - QPS Bio-Kinetic Clinical Applications (Patient Screening Only), Springfield, Missouri
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Methodist Physicians Clinic/CCT Research, Fremont, Nebraska
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Papillion Research Center/CCT Research, Papillion, Nebraska
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada / CCT Research, Las Vegas, Nevada
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - David Jurist Research Building, Hackensack, New Jersey
  - Hackensack University Medical Center Medical Plaza, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Velocity Clinical Research, Albuquerque, Albuquerque, New Mexico
  - Smith Allergy & Asthma Specialists, Horseheads, New York
  - NYU Langone Health, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - Accellacare - Cary, Cary, North Carolina
  - Accellacare - Charlotte, Charlotte, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare - Rocky Mount, Rocky Mount, North Carolina
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Plains Clinical Research Center, Fargo, North Dakota
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Senders Pediatrics, Cleveland, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - WellNow Urgent Care & Research, Dayton, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Tekton Research, LLC., Edmond, Oklahoma
  - Tekton Research, LLC., Moore, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tekton Research, LLC., Yukon, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Kaiser Permanente Northwest Center for Health Research, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Pharmacorp Clinical Trials, Charleston, South Carolina
  - Velocity Clinical Research, Columbia, Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Main Street Physician's Care, Little River, South Carolina
  - Clinical Trials of South Carolina, Moncks Corner, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - Velocity Clinical Research, Union, Union, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, Bristol, Tennessee
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Elligo Clinical Research Center, Austin, Texas
  - Benchmark Research, Austin, Texas
  - Tekton Research, LLC., Austin, Texas
  - Orion Clinical Research, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Headlands Research - Brownsville, Brownsville, Texas
  - WR-Global Medical Research, LLC, Dallas, Texas
  - DFW Clinical Research, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A, Dallas, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Proactive Clinical Research, LLC, Edinburg, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Family Care, Fort Worth, Texas
  - Allure Health, Friendswood, Texas
  - Trio Clinical Trials, Houston, Texas
  - Juno Research, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - Santa Clara Family Clinic, Houston, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Humble, Texas
  - Andres Garcia Zuniga, M.D., P.A., Laredo, Texas
  - SMS Clinical Research, Mesquite, Texas
  - AIM Trials, LLC, Plano, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Tekton Research, LLC., San Antonio, Texas
  - Javara - Privia Medical Group North Texas - Stephenville, Stephenville, Texas
  - Sugar Lakes Family Practice, PA, Sugar Land, Texas
  - DM Clinical Research, Martin Diagnostic Clinic, Tomball, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Crossroads Clinical Research, Victoria, Texas
  - Cope Family Medicine / CCT Research, Bountiful, Utah
  - South Ogden Family Medicine/ CCT Research, Ogden, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - Olympus Family Medicine/CCT Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Springville Dermatology - Springville/CCT Research, Springville, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Clinical Alliance for Research and Education - Infectious Diseases (CARE-ID), LLC, Annandale, Virginia
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia
  - Meridian Clinical Research LLC, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Centricity Research Suffolk Primary Care, Suffolk, Virginia
  - EvergreenHealth Medical Center, Kirkland, Washington
  - EvergreenHealth, Kirkland, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Kaiser Permanente Washington Health Research Institute (KPWHRI), Seattle, Washington
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
  - Seattle Clinical Research Center, Seattle, Washington
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Argentina (3):
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires
- Chile (3):
  - Enroll SpA, Santiago, Santiago Metropolitan
  - Centro Skin Med Limitada, Santiago, Santiago Metropolitan
  - CECIM, Santiago, Santiago Metropolitan
- New Zealand (11):
  - Pacific Clinical Research Network - Rotorua, Rotorua, Bay of Plenty
  - P3 Research - Tauranga, Tauranga, Bay of Plenty
  - Pacific Clinical Research Network - Forte, Christchurch, Canterbury
  - P3 Research - Hawke's Bay, Hastings, Hawke's Bay Region
  - Lakeland Clinical Trials Waikato, Hamilton, Waikato Region
  - Lakeland Clinical Trials Wellington, Upper Hutt, Wellington Region
  - Southern Clinical Trials Totara, Auckland
  - Optimal Clinical Trials North, Auckland
  - Optimal Clinical Trials, Auckland
  - Southern Clinical Trials Tasman, Nelson
  - P3 Research - Wellington, Wellington
- Philippines (12):
  - West Visayas State University Medical Center, Iloilo City, Iloilo
  - Tropical Disease Foundation, Makati City, National Capital Region
  - Health Cube Medical Clinics, Mandaluyong, National Capital Region
  - Mary Johnston Hospital, Manila, National Capital Region
  - Lung Center of the Philippines, Quezon City, National Capital Region
  - Far Eastern University Nicanor Reyes Medical Foundation, Quezon City, National Capital Region
  - Adventist Hospital Palawan, Puerto Princesa City, Palawan
  - De La Salle Medical and Health Sciences Institute, Dasmariñas
  - De La Salle Health Sciences Institute, Dasmariñas
  - Iloilo Doctors' Hospital, Iloilo City
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City
  - Philippine General Hospital, Manila
- South Africa (29):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Iatros International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - REIMED Reiger Park, Boksburg, Gauteng
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - Clinresco Centres, Kempton Park, Gauteng
  - Ubuntu Clinical Research - Krugersdorp, Krugersdorp, Gauteng
  - Ubuntu Clinical Research - Lenasia, Lenasia, Gauteng
  - Zinakekele Medicall Centre, Moloto, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Setshaba Research Centre, Pretoria, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Jongaie Research, Pretoria West, Gauteng
  - Wits Clinical Research, Soweto, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Val de Grace, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - Precise Clinical Solutions, Chatsworth, KwaZulu-Natal
  - Private Practice - Dr. Peter Sebastian, Chatsworth, KwaZulu-Natal
  - Synapta Clinical Research Centre, Durban, KwaZulu-Natal
  - MERCLINCO Middleburg, Middelburg, Mpumalanga
  - Aurum Institute - Rustenburg, Rustenburg, North West
  - TREAD Research (Pty)Ltd, Cape Town, Western Cape
  - TASK Applied Science, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - TREAD Research, Cape Town, Western Cape
  - Umzimkhulu Research Centre, uMzimkhulu

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fitz-Patrick D, McVinnie DS, Jackson LA, Crowther G, Geevarughese A, Cannon KD, Garcia LM, Pineiro Puebla Y, Yi Z, Cunliffe L, Maniar A, Zareba AM, Ianos CA, Gomme E, Koury K, Suphaphiphat Allen P, Anderson AS, Gurtman A, Lindert K; Pfizer C4781004 Trial Investigators. Efficacy, Immunogenicity, and Safety of Modified mRNA Influenza Vaccine. N Engl J Med. 2025 Nov 20;393(20):2001-2011. doi: 10.1056/NEJMoa2416779. PMID 41259756
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4781004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from northern hemisphere 2022-2023 and southern hemisphere 2023 were to be enrolled during respective influenza seasons and were stratified into 2 age groups: 18 to 64 years and more than or equal to (>=) 65 years.
Groups:
- qIRV: 18-64 Years: Participants aged 18-64 years were randomized to receive a single dose of quadrivalent influenza modified ribonucleic acid (modRNA) vaccine (qIRV) dose level 1 (low) intramuscularly (IM) on Day 1.
- Licensed QIV: 18-64 Years: Participants aged 18-64 years were randomized to receive a single dose of seasonal licensed quadrivalent influenza vaccine (QIV) IM per investigational product manual (IPM) on Day 1.
- qIRV: >=65 Years: Participants aged >=65 years were randomized to receive a single dose of qIRV dose level 2 (high) IM on Day 1.
- Licensed QIV: >=65 Years: Participants aged >=65 years were randomized to receive a single dose of seasonal licensed QIV IM per IPM on Day 1.
Period: Overall Study
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years | qIRV: >=65 Years | Licensed QIV: >=65 Years
Started | 9247 | 9251 | 13635 | 13656
Safety Set (Includes all randomized participants who received any study intervention at the specified dose level. Participants were included in the vaccination group corresponding to the study intervention that they actually received.) | 9191 | 9197 | 13557 | 13611
Completed | 8527 | 8598 | 13026 | 13043
Not Completed | 720 | 653 | 609 | 613
Not completed — Adverse Event | 1 | 0 | 2 | 5
Not completed — Lost to Follow-up | 487 | 427 | 146 | 166
Not completed — Physician Decision | 11 | 19 | 8 | 13
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 9 | 7
Not completed — Withdrawal by Subject | 168 | 134 | 331 | 322
Not completed — Death | 7 | 9 | 49 | 46
Not completed — Not vaccinated | 34 | 53 | 57 | 50
Not completed — No longer meets eligibility criteria | 0 | 0 | 3 | 2
Not completed — Other (Unspecified) | 8 | 10 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received the study intervention at the specified dose level. Participants were included in the vaccination group corresponding to the study intervention that they actually received.
Groups:
- qIRV: 18-64 Years: Participants aged 18-64 years were randomized to receive a single dose of modRNA qIRV dose level 1 (low) IM on Day 1.
- Licensed QIV: 18-64 Years: Participants aged 18-64 years were randomized to receive a single dose of seasonal licensed QIV IM per IPM on Day 1.
- Total: Total of all reporting groups
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years | qIRV: >=65 Years | Licensed QIV: >=65 Years | Total
Number analyzed (Participants) | 9191 | 9197 | 13557 | 13611 | 45556
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (13.05) | 43.1 (13.07) | 70.9 (4.91) | 70.8 (4.84) | 59.6 (16.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5395 | 5293 | 7649 | 7665 | 26002
  Male | 3796 | 3904 | 5908 | 5946 | 19554
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1961 | 1955 | 2041 | 2094 | 8051
  Not Hispanic or Latino | 7152 | 7156 | 11409 | 11430 | 37147
  Unknown or Not Reported | 78 | 86 | 107 | 87 | 358
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 73 | 69 | 37 | 42 | 221
  Asian | 372 | 350 | 1657 | 1691 | 4070
  Native Hawaiian or Other Pacific Islander | 24 | 32 | 64 | 70 | 190
  Black or African American | 1734 | 1753 | 2567 | 2562 | 8616
  White | 6780 | 6759 | 8974 | 8992 | 31505
  More than one race | 67 | 88 | 58 | 60 | 273
  Unknown or Not Reported | 141 | 146 | 200 | 194 | 681

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated Per-Protocol ILI Caused by Any Strain at Least 14 Days After Vaccination: 18-64 Years
Description: LCI was defined as influenza infection confirmed through through reverse transcription- polymerase chain reaction (RT-PCR) or culture at the central laboratory, unless otherwise specified. Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptoms concurrently with at least 1 systemic symptoms. Data was obtained during the 2022-2023 northern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population included all participants who were eligible, received the study intervention to which they were randomized, and had no important protocol deviations, with surveillance starting at least 14 days after vaccination.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.63 | 0.95
Statistical Analysis 1: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; Test type: Other; RVE = 34.5, 95% CI 2-sided [7.4 to 53.9]

2. Primary Outcome: Percentage of Participants Reporting First Episode of Laboratory-Confirmed Influenza (LCI) Cases With Associated Per-Protocol Influenza-Like Illness (ILI) Caused by Any Strain at Least 14 Days After Vaccination: >= 65 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptoms concurrently with at least 1 systemic symptoms. Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.59 | 0.56
Statistical Analysis 1: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; Test type: Other; RVE = -5.8, 95% CI 2-sided [-47.2 to 23.8]

3. Primary Outcome: Percentage of Participants Reporting Any Local Reactions Within 7 Days After Study Vaccination: 18-64 Years
Description: Local reactions included redness, swelling and pain at the injection site and were recorded by participants in an e-diary. All local reactions were graded based on Center for Biologics Evaluation and Research (CBER) toxicity guidelines as Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe) and Grade 4 (potentially life-threatening). In this outcome measure data is reported for any local reaction and any grade.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Reactogenicity e-diary safety included all participants who received the study intervention and had at least 1 day of e-diary data transferred for reactogenicity.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 3060 | 3067
Percentage of participants | 70.1 [68.5 to 71.7] | 43.1 [41.3 to 44.9]

4. Primary Outcome: Percentage of Participants Reporting Any Local Reactions Within 7 Days After Study Vaccination: >=65 Years
Description: as for outcome 3
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Reactogenicity e-diary safety set analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 3563 | 3563
Percentage of participants | 68.7 [67.2 to 70.3] | 25.8 [24.4 to 27.3]

5. Primary Outcome: Percentage of Participants Reporting Any Systemic Events Within 7 Days After Study Vaccination: 18-64 Years
Description: Systemic events (vomiting, diarrhoea, headache, Fatigue/tiredness, chills, new or worsened muscle pain and joint pain) were recorded by participants in an e-diary. All systemic events were graded based on CBER toxicity guidelines as Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe) and Grade 4 (potentially life-threatening). In this outcome measure data is reported for any systemic reaction and any grade.
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Reactogenicity e-diary safety set analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 3060 | 3067
Percentage of participants | 65.8 [64.0 to 67.4] | 48.7 [46.9 to 50.5]

6. Primary Outcome: Percentage of Participants Reporting Any Systemic Events Within 7 Days After Study Vaccination: >=65 Years
Description: as for outcome 5
Time Frame: From Day 1 to Day 7 after study vaccination
Population: Reactogenicity e-diary safety set analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 3563 | 3563
Percentage of participants | 58.6 [57.0 to 60.2] | 34.9 [33.3 to 36.4]

7. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) From Study Vaccination Through 4 Weeks After Study Vaccination: 18-64 Years
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Results excluded local reactions and systemic events data.
Time Frame: From study vaccination on Day 1 through 4 weeks after study vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9191 | 9197
Percentage of participants | 6.7 [6.2 to 7.3] | 4.9 [4.5 to 5.4]

8. Primary Outcome: Percentage of Participants Reporting AEs From Study Vaccination Through 4 Weeks After Study Vaccination: >=65 Years
Description: as for outcome 7
Time Frame: From study vaccination on Day 1 through 4 weeks after study vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13557 | 13611
Percentage of participants | 8.7 [8.2 to 9.1] | 5.9 [5.5 to 6.3]

9. Primary Outcome: Percentage of Participants Reporting AEs From Study Vaccination Through 4 Weeks After Study Vaccination: >=18 Years
Description: as for outcome 7
Time Frame: From study vaccination on Day 1 through 4 weeks after study vaccination
Population: Analysis population included all participants who received the study intervention. Data was planned to be analyzed in participants aged >=18 years (combined for 18-64 years and >65 years) as pre-specified in the protocol. The analysis includes participants who received qIRV at either dose level, as well as QIV.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- qIRV (>=18 Years): Participants aged >=18 years were randomized to receive a single dose of qIRV dose level 1 (low) and dose level 2 (high) IM on Day 1.
- Licensed QIV (>=18 Years): Participants aged >=65 years were randomized to receive a single dose of seasonal licensed QIV IM per IPM on Day 1.
Arm/Group | qIRV (>=18 Years) | Licensed QIV (>=18 Years)
Number analyzed (Participants) | 22787 | 22808
Percentage of participants | 7.9 [7.5 to 8.2] | 5.5 [5.2 to 5.8]

10. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) From Study Vaccination Through 6 Months After Study Vaccination: 18-64 Years
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect.
Time Frame: From Day 1 up to 6 months after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9191 | 9197
Percentage of participants | 0.9 [0.7 to 1.1] | 1.0 [0.8 to 1.2]

11. Primary Outcome: Percentage of Participants Reporting SAEs From Study Vaccination Through 6 Months After Study Vaccination: >=65 Years
Description: as for outcome 10
Time Frame: From Day 1 up to 6 months after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13557 | 13611
Percentage of participants | 2.3 [2.1 to 2.6] | 2.2 [1.9 to 2.4]

12. Primary Outcome: Percentage of Participants Reporting SAEs From Study Vaccination Through 6 Months After Study Vaccination: >=18 Years
Description: as for outcome 10
Time Frame: From Day 1 up to 6 months after vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV (>=18 Years) | Licensed QIV (>=18 Years)
Number analyzed (Participants) | 22787 | 22808
Percentage of participants | 1.8 [1.6 to 1.9] | 1.7 [1.5 to 1.9]

13. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated Per-Protocol ILI Caused by All Matched Strains at Least 14 Days After Vaccination: 18-64 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. Data was obtained during the 2022-2023 northern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.23 | 0.34

14. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated Per-Protocol ILI Caused by All Matched Strains at Least 14 Days After Vaccination: >=65 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.34 | 0.36

15. Secondary Outcome: Percentage of Participants Reporting First Episode of Culture Confirmed Influenza (CCI) With Associated Per-Protocol ILI Caused by Any Strain at Least 14 Days After Vaccination: 18-64 Years
Description: CCI was defined as influenza infection confirmed through culture at the central laboratory, unless otherwise specified. Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptom concurrently with at least 1 systemic symptom. Data was obtained during the 2022-2023 northern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.23 | 0.34

16. Secondary Outcome: Percentage of Participants Reporting First Episode of CCI With Associated Per-Protocol ILI Caused by Any Strain at Least 14 Days After Vaccination: >=65 Years
Description: CCI was defined as influenza infection confirmed through culture at the central laboratory, unless otherwise specified. Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptom concurrently with at least 1 systemic symptom. Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.34 | 0.36

17. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated ILI as Defined by Modified Centers for Disease Control and Prevention (CDC) Caused by Any Strain at Least 14 Days After Vaccination: 18-64 Years
Description: as for outcome 13
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.46 | 0.61

18. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated ILI as Defined by Modified CDC Caused by Any Strain at Least 14 Days After Vaccination: >=65 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. ILI defined modified CDC: occurrence (new onset or worsening of preexisting condition) of at least 1 of the following respiratory symptoms concurrently with an oral temperature >37.2 deg C (>99.0 deg F), sore throat or cough. Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.36 | 0.30

19. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated ILI as Defined by World Health Organization (WHO) Caused by Any Strain at Least 14 Days After Vaccination: 18-64 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. ILI as per WHO was defined as occurrence (new onset or worsening of preexisting condition) of a cough concurrently with an oral temperature >=38.0 deg C (>= 100.4 deg F). Data was obtained during the 2022-2023 northern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.27 | 0.35

20. Secondary Outcome: Percentage of Participants Reporting First Episode of LCI Cases With Associated ILI as Defined by WHO Caused by Any Strain at Least 14 Days After Vaccination: >=65 Years
Description: LCI was defined as influenza infection confirmed through RT-PCR or culture at the central laboratory, unless otherwise specified. ILI as per WHO was defined as occurrence (new onset or worsening of preexisting condition) of a cough concurrently with an oral temperature >=38.0 deg C (>= 100.4 deg F). Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.23 | 0.22

21. Secondary Outcome: Percentage of Participants Reporting First Episode Cases of Influenza as Confirmed by RT-PCR or Local RT-PCR or Culture, With Associated Per-Protocol ILI at Least 14 Days After Vaccination: 18-64 Years
Description: Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptom concurrently with at least 1 systemic symptom. Data was obtained during the 2022-2023 northern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 to surveillance cut-off (approximately 6 months)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 9118 | 9120
Percentage of participants | 0.66 | 0.98

22. Secondary Outcome: Percentage of Participants Reporting First Episode Cases of Influenza as Confirmed by Central RT-PCR or Local RT-PCR or Culture, With Associated Per-Protocol ILI at Least 14 Days After Vaccination: >=65 Years
Description: Per-protocol ILI was defined as occurrence (new onset or worsening of preexisting condition) of at least 1 respiratory symptom concurrently with at least 1 systemic symptom. Data was obtained during the 2022-2023 northern and southern hemisphere influenza season up to surveillance cut-off decided by Sponsor.
Time Frame: Day 15 up to primary surveillance cut-off (approximately 1 year)
Population: Evaluable efficacy population analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 13392 | 13456
Percentage of participants | 0.65 | 0.62

23. Secondary Outcome: HAI GMTs Used to Determine GMRs of qIRV to Licensed QIV at 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: 18-64 Years
Description: Geometric mean titers (GMTs) and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the student t distribution) and were reported in the descriptive section. Geometric mean ratios (GMRs) were estimated by the ratio of the GMTs between qIRV recipients compared to licensed QIV recipients vaccine groups and were reported in the statistical analysis section.
Time Frame: 4 Weeks after vaccination
Population: Evaluable immunogenicity set (Based on HAI Assay 2): eligible participants, received study intervention to which they were randomized, had blood drawn for assay testing within specified time frame, had at least 1 valid, determinate assay result (HAIs determinate assay 2) at 4-week postvaccination, no important protocol deviations. All participants reported under "N" contributed data to table but may not have evaluable data for every row. "n"=number of participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 739 | 746
Titers
  A/H3N2: number analyzed (Participants) | 738 | 746
  A/H3N2 | 222.3 [206.0 to 240.0] | 180.4 [166.6 to 195.4]
  A/H1N1: number analyzed (Participants) | 738 | 746
  A/H1N1 | 397.7 [367.8 to 430.0] | 321.7 [294.6 to 351.2]
  B/Yamagata: number analyzed (Participants) | 736 | 743
  B/Yamagata | 84.5 [79.4 to 90.0] | 115.9 [108.5 to 123.8]
  B/Victoria: number analyzed (Participants) | 734 | 736
  B/Victoria | 21.3 [19.3 to 23.6] | 70.6 [63.6 to 78.4]
Statistical Analysis 1: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H3N2; Test type: Other; GMR = 1.23, 95% CI 2-sided [1.10 to 1.38]
Statistical Analysis 2: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H1N1; Test type: Other; GMR = 1.24, 95% CI 2-sided [1.10 to 1.39]
Statistical Analysis 3: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Yamagata; Test type: Other; GMR = 0.73, 95% CI 2-sided [0.67 to 0.80]
Statistical Analysis 4: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Victoria; Test type: Other; GMR = 0.3, 95% CI 2-sided [0.26 to 0.35]

24. Secondary Outcome: HAI GMTs Used to Determine GMRs of qIRV to Licensed QIV for 2022-2023 Northern Hemisphere at 4 Weeks After Vaccination- Based on HAI Assay 2: >=65 Years
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the student t distribution) and were reported in the descriptive section. GMRs were estimated by the ratio of the GMTs between qIRV recipients compared to licensed QIV recipients vaccine groups and were reported in the statistical analysis section.
Time Frame: 4 Weeks after vaccination
Population: Evaluable immunogenicity set (Based on HAI Assay 2) analyzed. All participants reported under "Number of Participants Analyzed" contributed data to the table but may not have evaluable data for every row. Here, "Number analyzed" signifies number of participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 754 | 740
Titers
  A/H3N2: number analyzed (Participants) | 753 | 738
  A/H3N2 | 296.0 [273.7 to 320.1] | 179.8 [166.3 to 194.5]
  A/H1N1: number analyzed (Participants) | 754 | 733
  A/H1N1 | 240.0 [220.3 to 261.3] | 140.6 [129.2 to 152.9]
  B/Yamagata: number analyzed (Participants) | 749 | 732
  B/Yamagata | 57.6 [54.1 to 61.2] | 55.3 [52.0 to 58.9]
  B/Victoria: number analyzed (Participants) | 750 | 734
  B/Victoria | 82.1 [75.0 to 89.9] | 134.8 [123.5 to 147.3]
Statistical Analysis 1: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H3N2; Test type: Other; GMR = 1.65, 95% CI 2-sided [1.47 to 1.84]
Statistical Analysis 2: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H1N1; Test type: Other; GMR = 1.71, 95% CI 2-sided [1.51 to 1.92]
Statistical Analysis 3: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Yamagata; Test type: Other; GMR = 1.04, 95% CI 2-sided [0.95 to 1.14]
Statistical Analysis 4: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Victoria; Test type: Other; GMR = 0.61, 95% CI 2-sided [0.54 to 0.69]

25. Secondary Outcome: Percentage of Participants and Difference in Percentage of Participants Achieving Seroconversion at 4 Weeks After Vaccination With qIRV and Licensed QIV for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: 18-64 Years
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Percentage of participants achieving seroconversion for each strain at 4 weeks after vaccination and exact 2-sided 95% CI is presented in the descriptive section. Difference in percentage of participants (qIRV - QIV) achieving HAI seroconversion for each strain at 4 weeks after vaccination is presented in the statistical analysis section.
Time Frame: 4 Weeks after vaccination
Population: Evaluable immunogenicity set (Based on HAI Assay 2) analyzed. Here, Participants reported under "Number of Participants Analyzed" contributed data but may not be evaluable for every row and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 739 | 746
Percentage of Participants
  A/H3N2: number analyzed (Participants) | 735 | 746
  A/H3N2 | 64.2 [60.6 to 67.7] | 52.8 [49.2 to 56.4]
  A/H1N1: number analyzed (Participants) | 735 | 743
  A/H1N1 | 66.1 [62.6 to 69.5] | 52.5 [48.8 to 56.1]
  B/Yamagata: number analyzed (Participants) | 736 | 743
  B/Yamagata | 13.9 [11.4 to 16.6] | 29.2 [26.0 to 32.6]
  B/Victoria: number analyzed (Participants) | 731 | 733
  B/Victoria | 11.4 [9.1 to 13.9] | 51.8 [48.2 to 55.5]
Statistical Analysis 1: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H3N2: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = 11.4, 95% CI 2-sided [6.4 to 16.4]
Statistical Analysis 2: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H1N1: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = 13.6, 95% CI 2-sided [8.6 to 18.6]
Statistical Analysis 3: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Yamagata: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = -15.3, 95% CI 2-sided [-19.5 to -11.2]
Statistical Analysis 4: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Victoria: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = -40.5, 95% CI 2-sided [-44.7 to -36.1]

26. Secondary Outcome: Percentage of Participants and Difference in Percentage of Participants Achieving Seroconversion at 4 Weeks After Vaccination With qIRV and Licensed QIV for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: >=65 Years
Description: as for outcome 25
Time Frame: 4 Weeks after vaccination
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 754 | 740
Percentage of participants
  A/H3N2: number analyzed (Participants) | 748 | 735
  A/H3N2 | 53.2 [49.6 to 56.8] | 31.6 [28.2 to 35.1]
  A/H1N1: number analyzed (Participants) | 749 | 730
  A/H1N1 | 50.2 [46.6 to 53.8] | 24.5 [21.4 to 27.8]
  B/Yamagata: number analyzed (Participants) | 747 | 731
  B/Yamagata | 6.4 [4.8 to 8.4] | 8.5 [6.6 to 10.7]
  B/Victoria: number analyzed (Participants) | 750 | 731
  B/Victoria | 10.9 [8.8 to 13.4] | 33.5 [30.1 to 37.1]
Statistical Analysis 1: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H3N2: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = 21.6, 95% CI 2-sided [16.7 to 26.5]
Statistical Analysis 2: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H1N1: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = 25.7, 95% CI 2-sided [20.9 to 30.4]
Statistical Analysis 3: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Yamagata: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = -2.1, 95% CI 2-sided [-4.8 to 0.6]
Statistical Analysis 4: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Victoria: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in percentage = -22.6, 95% CI 2-sided [-26.7 to -18.5]

27. Secondary Outcome: HAI GMTs Used to Determine GMRs of qIRV to Licensed QIV for 2022-2023 Northern Hemisphere at 4 Weeks After Vaccination- Based on HAI Assay 1: 18-64 Years
Description: GMTs and 2-sided 95% CIs were reported in the descriptive section. GMRs were estimated by the ratio of the GMTs between qIRV recipients compared to licensed QIV recipients vaccine groups and were reported in the statistical analysis section.
Time Frame: 4 Weeks after vaccination
Population: Evaluable immunogenicity set (Based on HAI Assay 1) analyzed. Participants reported under "Number of Participants Analyzed" contributed data but may not be evaluable for every row. "Number Analyzed": participants evaluable for rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 1867 | 1871
Titers
  A/H3N2: number analyzed (Participants) | 1837 | 1840
  A/H3N2 | 117.3 [111.2 to 123.6] | 61.1 [57.8 to 64.5]
  A/H1N1: number analyzed (Participants) | 1864 | 1863
  A/H1N1 | 203.7 [193.3 to 214.8] | 121.2 [114.1 to 128.8]
  B/Yamagata: number analyzed (Participants) | 1864 | 1864
  B/Yamagata | 55.0 [52.6 to 57.5] | 62.4 [59.4 to 65.5]
  B/Victoria: number analyzed (Participants) | 1866 | 1868
  B/Victoria | 16.7 [15.8 to 17.6] | 28.7 [27.0 to 30.6]
Statistical Analysis 1: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H3N2; Test type: Other; GMR = 1.92, 95% CI 2-sided [1.78 to 2.07]
Statistical Analysis 2: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H1N1; Test type: Other; GMR = 1.68, 95% CI 2-sided [1.55 to 1.82]
Statistical Analysis 3: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Yamagata; Test type: Other; GMR = 0.88, 95% CI 2-sided [0.82 to 0.94]
Statistical Analysis 4: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Victoria; Test type: Other; GMR = 0.58, 95% CI 2-sided [0.53 to 0.63]

28. Secondary Outcome: HAI GMTs Used to Determine GMRs of qIRV to Licensed QIV for 2022-2023 Northern Hemisphere at 4 Weeks After Vaccination - Based on HAI Assay 1: >=65 Years
Description: as for outcome 27
Time Frame: 4 Weeks after vaccination
Population: Evaluable immunogenicity set (Based on HAI Assay 1) analyzed. Participants reported under "Number of Participants Analyzed" contributed data but may not be evaluable for every row. "Number Analyzed" signifies participants evaluable for rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 2447 | 2441
Titers
  A/H3N2: number analyzed (Participants) | 2431 | 2420
  A/H3N2 | 98.2 [93.9 to 102.8] | 41.3 [39.4 to 43.3]
  A/H1N1: number analyzed (Participants) | 2443 | 2433
  A/H1N1 | 131.8 [125.9 to 138.0] | 55.6 [52.8 to 58.5]
  B/Yamagata: number analyzed (Participants) | 2440 | 2433
  B/Yamagata | 38.9 [37.5 to 40.3] | 28.6 [27.6 to 29.7]
  B/Victoria: number analyzed (Participants) | 2446 | 2436
  B/Victoria | 40.1 [38.4 to 41.8] | 52.9 [50.4 to 55.5]
Statistical Analysis 1: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H3N2; Test type: Other; GMR = 2.38, 95% CI 2-sided [2.23 to 2.54]
Statistical Analysis 2: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H1N1; Test type: Other; GMR = 2.37, 95% CI 2-sided [2.22 to 2.54]
Statistical Analysis 3: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Yamagata; Test type: Other; GMR = 1.36, 95% CI 2-sided [1.29 to 1.43]
Statistical Analysis 4: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Victoria; Test type: Other; GMR = 0.76, 95% CI 2-sided [0.71 to 0.81]

29. Secondary Outcome: Percentage of Participants and Difference in Percentage of Participants Achieving Seroconversion at 4 Weeks After Vaccination With qIRV and Licensed QIV for 2022-2023 Northern Hemisphere-Based on HAI Assay 1: 18-64 Years
Description: as for outcome 25
Time Frame: 4 Weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 1867 | 1871
Percentage of participants
  A/H3N2: number analyzed (Participants) | 1807 | 1808
  A/H3N2 | 73.1 [71.0 to 75.1] | 46.3 [44.0 to 48.6]
  A/H1N1: number analyzed (Participants) | 1833 | 1831
  A/H1N1 | 78.3 [76.4 to 80.2] | 51.4 [49.1 to 53.8]
  B/Yamagata: number analyzed (Participants) | 1833 | 1832
  B/Yamagata | 30.0 [27.9 to 32.1] | 33.5 [31.4 to 35.7]
  B/Victoria: number analyzed (Participants) | 1835 | 1836
  B/Victoria | 13.5 [12.0 to 15.2] | 32.7 [30.6 to 34.9]
Statistical Analysis 1: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H3N2: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = 26.8, 95% CI 2-sided [23.7 to 29.9]
Statistical Analysis 2: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; A/H1N1: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = 26.9, 95% CI 2-sided [23.9 to 29.8]
Statistical Analysis 3: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Yamagata: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = -3.6, 95% CI 2-sided [-6.6 to -0.6]
Statistical Analysis 4: Comparison: qIRV: 18-64 Years vs Licensed QIV: 18-64 Years; B/Victoria: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = -19.2, 95% CI 2-sided [-21.9 to -16.6]

30. Secondary Outcome: Percentage of Participants and Difference in Percentage of Participants Achieving Seroconversion at 4 Weeks After Vaccination With qIRV and Licensed QIV for 2022-2023 Northern Hemisphere- Based on HAI Assay 1: >=65 Years
Description: as for outcome 25
Time Frame: 4 Weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 2447 | 2441
Percentage of participants
  A/H3N2: number analyzed (Participants) | 2336 | 2331
  A/H3N2 | 66.0 [64.0 to 67.9] | 28.1 [26.3 to 30.0]
  A/H1N1: number analyzed (Participants) | 2348 | 2344
  A/H1N1 | 68.4 [66.5 to 70.3] | 23.5 [21.8 to 25.2]
  B/Yamagata: number analyzed (Participants) | 2345 | 2344
  B/Yamagata | 22.6 [21.0 to 24.4] | 12.0 [10.7 to 13.4]
  B/Victoria: number analyzed (Participants) | 2351 | 2347
  B/Victoria | 19.8 [18.2 to 21.4] | 33.6 [31.7 to 35.5]
Statistical Analysis 1: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H3N2: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = 37.9, 95% CI 2-sided [35.2 to 40.5]
Statistical Analysis 2: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; A/H1N1: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = 44.9, 95% CI 2-sided [42.4 to 47.4]
Statistical Analysis 3: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Yamagata: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = 10.6, 95% CI 2-sided [8.5 to 12.8]
Statistical Analysis 4: Comparison: qIRV: >=65 Years vs Licensed QIV: >=65 Years; B/Victoria: 2-Sided CI, difference in percents (qIRV - Licensed QIV), expressed as a percentage; Test type: Other; Difference in Percentage = -13.8, 95% CI 2-sided [-16.3 to -11.3]

31. Secondary Outcome: HAI GMTs at Baseline for the 2022-2023 Northern Hemisphere - Based on HAI Assay 2: 18-64 Years
Time Frame: Baseline (Before Vaccination)
Population: Evaluable immunogenicity set (Based on HAI Assay 2) analyzed. Participants reported under "Number of Participants Analyzed" contributed data but may not be evaluable for every row. "Number Analyzed": participants evaluable for rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 739 | 746
Titers
  A/H3N2: number analyzed (Participants) | 735 | 746
  A/H3N2 | 42.9 [39.7 to 46.3] | 42.3 [39.3 to 45.4]
  A/H1N1: number analyzed (Participants) | 735 | 743
  A/H1N1 | 58.0 [51.8 to 64.9] | 50.5 [45.2 to 56.4]
  B/Yamagata: number analyzed (Participants) | 736 | 743
  B/Yamagata | 49.2 [45.9 to 52.8] | 46.2 [43.0 to 49.6]
  B/Victoria: number analyzed (Participants) | 732 | 737
  B/Victoria | 13.0 [11.9 to 14.2] | 13.5 [12.4 to 14.8]

32. Secondary Outcome: HAI GMTs at Baseline for 2022-2023 Northern Hemisphere - Based on HAI Assay 2: >=65 Years
Time Frame: Baseline (Before Vaccination)
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 754 | 740
Titers
  A/H3N2: number analyzed (Participants) | 748 | 735
  A/H3N2 | 71.2 [67.1 to 75.6] | 68.6 [64.7 to 72.7]
  A/H1N1: number analyzed (Participants) | 749 | 731
  A/H1N1 | 60.2 [54.4 to 66.6] | 58.3 [52.8 to 64.4]
  B/Yamagata: number analyzed (Participants) | 749 | 731
  B/Yamagata | 38.7 [36.5 to 41.1] | 36.8 [34.5 to 39.2]
  B/Victoria: number analyzed (Participants) | 751 | 731
  B/Victoria | 47.5 [43.3 to 52.2] | 43.5 [39.4 to 48.0]

33. Secondary Outcome: HAI Geometric Mean Fold Rise (GMFR) From Before Vaccination to 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: 18-64 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination (baseline).
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 739 | 746
Fold rise
  A/H3N2: number analyzed (Participants) | 735 | 746
  A/H3N2 | 4.9 [4.5 to 5.2] | 4.1 [3.8 to 4.4]
  A/H1N1: number analyzed (Participants) | 735 | 743
  A/H1N1 | 6.0 [5.5 to 6.6] | 5.6 [5.0 to 6.2]
  B/Yamagata: number analyzed (Participants) | 736 | 743
  B/Yamagata | 1.7 [1.6 to 1.8] | 2.4 [2.2 to 2.5]
  B/Victoria: number analyzed (Participants) | 731 | 733
  B/Victoria | 1.4 [1.4 to 1.5] | 3.9 [3.6 to 4.2]

34. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: >=65 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination (baseline).
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 754 | 740
Fold rise
  A/H3N2: number analyzed (Participants) | 748 | 735
  A/H3N2 | 4.2 [3.9 to 4.4] | 2.6 [2.5 to 2.8]
  A/H1N1: number analyzed (Participants) | 749 | 730
  A/H1N1 | 3.7 [3.4 to 3.9] | 2.2 [2.0 to 2.4]
  B/Yamagata: number analyzed (Participants) | 747 | 731
  B/Yamagata | 1.4 [1.4 to 1.5] | 1.4 [1.4 to 1.5]
  B/Victoria: number analyzed (Participants) | 750 | 731
  B/Victoria | 1.6 [1.6 to 1.7] | 2.8 [2.6 to 3.0]

35. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 2: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 739 | 746
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 735 | 746
  Baseline: A/H3N2 | 65.0 [61.5 to 68.5] | 63.1 [59.6 to 66.6]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 738 | 746
  4 Weeks after vaccination: A/H3N2 | 99.2 [98.2 to 99.7] | 96.5 [94.9 to 97.7]
  Baseline: A/H1N1: number analyzed (Participants) | 735 | 743
  Baseline: A/H1N1 | 68.0 [64.5 to 71.4] | 63.5 [59.9 to 67.0]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 738 | 746
  4 Weeks after vaccination: A/H1N1 | 98.4 [97.2 to 99.2] | 96.6 [95.1 to 97.8]
  Baseline: B/Yamagata: number analyzed (Participants) | 736 | 743
  Baseline: B/Yamagata | 71.3 [67.9 to 74.6] | 69.3 [65.9 to 72.6]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 736 | 743
  4 Weeks after vaccination: B/Yamagata | 88.7 [86.2 to 90.9] | 93.0 [90.9 to 94.7]
  Baseline: B/Victoria: number analyzed (Participants) | 732 | 737
  Baseline: B/Victoria | 25.7 [22.6 to 29.0] | 24.6 [21.5 to 27.8]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 734 | 736
  4 Weeks after vaccination: B/Victoria | 38.6 [35.0 to 42.2] | 72.7 [69.3 to 75.9]

36. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere - Based on HAI Assay 2: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 754 | 740
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 748 | 735
  Baseline: A/H3N2 | 84.5 [81.7 to 87.0] | 85.6 [82.8 to 88.0]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 753 | 738
  4 Weeks after vaccination: A/H3N2 | 99.6 [98.8 to 99.9] | 97.3 [95.8 to 98.3]
  Baseline: A/H1N1: number analyzed (Participants) | 749 | 731
  Baseline: A/H1N1 | 70.5 [67.1 to 73.7] | 73.2 [69.8 to 76.4]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 754 | 733
  4 Weeks after vaccination: A/H1N1 | 96.2 [94.5 to 97.4] | 92.1 [89.9 to 93.9]
  Baseline: B/Yamagata: number analyzed (Participants) | 749 | 731
  Baseline: B/Yamagata | 60.9 [57.3 to 64.4] | 60.7 [57.1 to 64.3]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 749 | 732
  4 Weeks after vaccination: B/Yamagata | 77.3 [74.1 to 80.3] | 75.0 [71.7 to 78.1]
  Baseline: B/Victoria: number analyzed (Participants) | 751 | 731
  Baseline: B/Victoria | 64.4 [60.9 to 67.9] | 61.6 [57.9 to 65.1]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 750 | 734
  4 Weeks after vaccination: B/Victoria | 78.7 [75.6 to 81.5] | 89.8 [87.4 to 91.9]

37. Secondary Outcome: HAI GMTs at Baseline for 2022-2023 Northern Hemisphere - Based on HAI Assay 1: 18-64 Years
Time Frame: Baseline
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 1867 | 1871
Titers
  A/H3N2: number analyzed (Participants) | 1807 | 1808
  A/H3N2 | 18.2 [17.3 to 19.2] | 17.6 [16.7 to 18.5]
  A/H1N1: number analyzed (Participants) | 1833 | 1831
  A/H1N1 | 22.7 [21.4 to 24.1] | 23.1 [21.8 to 24.5]
  B/Yamagata: number analyzed (Participants) | 1833 | 1832
  B/Yamagata | 22.7 [21.6 to 23.8] | 22.7 [21.6 to 23.9]
  B/Victoria: number analyzed (Participants) | 1835 | 1836
  B/Victoria | 10.1 [9.6 to 10.6] | 10.1 [9.6 to 10.5]

38. Secondary Outcome: HAI GMTs at Baseline for 2022-2023 Northern Hemisphere- Based on HAI Assay 1: >=65 Years
Time Frame: Baseline
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 2447 | 2441
Titers
  A/H3N2: number analyzed (Participants) | 2336 | 2331
  A/H3N2 | 19.7 [18.9 to 20.6] | 19.0 [18.2 to 19.8]
  A/H1N1: number analyzed (Participants) | 2348 | 2344
  A/H1N1 | 25.2 [24.0 to 26.4] | 24.5 [23.4 to 25.8]
  B/Yamagata: number analyzed (Participants) | 2345 | 2344
  B/Yamagata | 18.1 [17.4 to 18.7] | 17.2 [16.6 to 17.8]
  B/Victoria: number analyzed (Participants) | 2351 | 2347
  B/Victoria | 20.0 [19.1 to 20.9] | 19.7 [18.8 to 20.6]

39. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 1: 18-64 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination (baseline).
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 1867 | 1871
Fold rise
  A/H3N2: number analyzed (Participants) | 1807 | 1808
  A/H3N2 | 5.4 [5.1 to 5.6] | 2.9 [2.8 to 3.1]
  A/H1N1: number analyzed (Participants) | 1833 | 1831
  A/H1N1 | 7.5 [7.1 to 7.9] | 4.4 [4.1 to 4.7]
  B/Yamagata: number analyzed (Participants) | 1833 | 1832
  B/Yamagata | 2.2 [2.1 to 2.2] | 2.4 [2.3 to 2.5]
  B/Victoria: number analyzed (Participants) | 1835 | 1836
  B/Victoria | 1.4 [1.4 to 1.5] | 2.2 [2.1 to 2.3]

40. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere- Based on HAI Assay 1: >=65 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination.
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 2447 | 2441
Fold rise
  A/H3N2: number analyzed (Participants) | 2336 | 2331
  A/H3N2 | 4.2 [4.1 to 4.4] | 1.9 [1.9 to 2.0]
  A/H1N1: number analyzed (Participants) | 2348 | 2344
  A/H1N1 | 4.5 [4.4 to 4.7] | 2.0 [1.9 to 2.1]
  B/Yamagata: number analyzed (Participants) | 2345 | 2344
  B/Yamagata | 1.9 [1.9 to 2.0] | 1.5 [1.5 to 1.5]
  B/Victoria: number analyzed (Participants) | 2351 | 2347
  B/Victoria | 1.8 [1.8 to 1.9] | 2.4 [2.3 to 2.5]

41. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere - Based on HAI Assay 1: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 1867 | 1871
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 1807 | 1808
  Baseline: A/H3N2 | 36.8 [34.6 to 39.1] | 35.2 [33.0 to 37.4]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 1837 | 1840
  4 Weeks after vaccination: A/H3N2 | 91.1 [89.7 to 92.4] | 75.8 [73.7 to 77.7]
  Baseline: A/H1N1: number analyzed (Participants) | 1833 | 1831
  Baseline: A/H1N1 | 41.6 [39.4 to 43.9] | 44.9 [42.7 to 47.3]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 1864 | 1863
  4 Weeks after vaccination: A/H1N1 | 95.0 [93.9 to 95.9] | 86.8 [85.2 to 88.3]
  Baseline: B/Yamagata: number analyzed (Participants) | 1833 | 1832
  Baseline: B/Yamagata | 42.2 [40.0 to 44.5] | 43.0 [40.7 to 45.3]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 1864 | 1864
  4 Weeks after vaccination: B/Yamagata | 75.3 [73.2 to 77.2] | 76.7 [74.7 to 78.6]
  Baseline: B/Victoria: number analyzed (Participants) | 1835 | 1836
  Baseline: B/Victoria | 16.3 [14.6 to 18.1] | 15.5 [13.8 to 17.2]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 1866 | 1868
  4 Weeks after vaccination: B/Victoria | 31.9 [29.8 to 34.1] | 47.0 [44.7 to 49.3]

42. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2022-2023 Northern Hemisphere - Based on HAI Assay 1: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 2447 | 2441
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 2336 | 2331
  Baseline: A/H3N2 | 40.4 [38.4 to 42.4] | 37.6 [35.6 to 39.6]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 2431 | 2420
  4 Weeks after vaccination: A/H3N2 | 88.3 [87.0 to 89.6] | 64.6 [62.7 to 66.5]
  Baseline: A/H1N1: number analyzed (Participants) | 2348 | 2344
  Baseline: A/H1N1 | 46.4 [44.4 to 48.5] | 44.4 [42.4 to 46.4]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 2443 | 2433
  4 Weeks after vaccination: A/H1N1 | 91.7 [90.6 to 92.8] | 70.6 [68.8 to 72.4]
  Baseline: B/Yamagata: number analyzed (Participants) | 2345 | 2344
  Baseline: B/Yamagata | 31.0 [29.1 to 32.9] | 28.3 [26.5 to 30.2]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 2440 | 2433
  4 Weeks after vaccination: B/Yamagata | 65.1 [63.2 to 67.0] | 50.2 [48.2 to 52.2]
  Baseline: B/Victoria: number analyzed (Participants) | 2351 | 2347
  Baseline: B/Victoria | 36.3 [34.3 to 38.3] | 35.2 [33.2 to 37.1]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 2446 | 2436
  4 Weeks after vaccination: B/Victoria | 63.6 [61.7 to 65.5] | 69.0 [67.1 to 70.8]

43. Secondary Outcome: HAI GMTs at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 2: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: As there was no participant from southern hemisphere aged 18-64 years, no data was collected for this outcome measure. Therefore, there was no analysis performed for this outcome measure.
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: HAI GMTs at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 2: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Titers
  Baseline: A/H3N2: number analyzed (Participants) | 386 | 386
  Baseline: A/H3N2 | 84.1 [77.1 to 91.8] | 82.9 [76.1 to 90.2]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 390 | 388
  4 Weeks after vaccination: A/H3N2 | 460.9 [414.8 to 512.0] | 272.2 [244.3 to 303.3]
  Baseline: A/H1N1: number analyzed (Participants) | 388 | 386
  Baseline: A/H1N1 | 10.9 [9.7 to 12.3] | 12.2 [10.8 to 13.8]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 390 | 389
  4 Weeks after vaccination: A/H1N1 | 73.8 [62.9 to 86.5] | 92.7 [80.0 to 107.4]
  Baseline: B/Yamagata: number analyzed (Participants) | 386 | 385
  Baseline: B/Yamagata | 35.5 [32.1 to 39.2] | 37.5 [33.8 to 41.5]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 387 | 389
  4 Weeks after vaccination: B/Yamagata | 70.0 [64.0 to 76.5] | 81.4 [74.5 to 88.9]
  Baseline: B/Victoria: number analyzed (Participants) | 385 | 382
  Baseline: B/Victoria | 34.0 [29.6 to 39.2] | 31.1 [26.9 to 36.0]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 386 | 382
  4 Weeks after vaccination: B/Victoria | 77.9 [69.1 to 87.8] | 124.2 [109.9 to 140.5]

45. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2023 Southern- Based on HAI Assay 2: 18-64 Years
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2023 Southern Hemisphere- Based on HAI Assay 2: >=65 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination (baseline).
Time Frame: Before vaccination (Baseline) to 4 weeks after vaccination
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Fold rise
  A/H3N2: number analyzed (Participants) | 386 | 385
  A/H3N2 | 5.5 [5.0 to 6.0] | 3.3 [3.0 to 3.6]
  A/H1N1: number analyzed (Participants) | 388 | 385
  A/H1N1 | 4.8 [4.2 to 5.4] | 5.4 [4.7 to 6.2]
  B/Yamagata: number analyzed (Participants) | 386 | 383
  B/Yamagata | 1.8 [1.7 to 2.0] | 2.0 [1.9 to 2.2]
  B/Victoria: number analyzed (Participants) | 385 | 379
  B/Victoria | 2.0 [1.9 to 2.2] | 3.3 [3.0 to 3.8]

47. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion at 4 Weeks After Vaccination for the 2023 Southern Hemisphere - Based on HAI Assay 2: 18-64 Years
Time Frame: 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion at 4 Weeks After Vaccination for 2023 Southern Hemisphere- Based on HAI Assay 2: >=65 Years
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest.
Time Frame: 4 weeks after vaccination
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Percentage of participants
  A/H3N2: number analyzed (Participants) | 386 | 385
  A/H3N2 | 68.9 [64.0 to 73.5] | 41.6 [36.6 to 46.7]
  A/H1N1: number analyzed (Participants) | 388 | 385
  A/H1N1 | 58.5 [53.4 to 63.5] | 58.7 [53.6 to 63.7]
  B/Yamagata: number analyzed (Participants) | 386 | 385
  B/Yamagata | 16.3 [12.8 to 20.4] | 21.6 [17.6 to 26.0]
  B/Victoria: number analyzed (Participants) | 385 | 379
  B/Victoria | 21.0 [17.1 to 25.5] | 36.4 [31.6 to 41.5]

49. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 2: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 2: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 386 | 386
  Baseline: A/H3N2 | 93.8 [90.9 to 96.0] | 94.0 [91.2 to 96.2]
  4 weeks after vaccination: A/H3N2: number analyzed (Participants) | 390 | 388
  4 weeks after vaccination: A/H3N2 | 100.0 [99.1 to 100.0] | 99.0 [97.4 to 99.7]
  Baseline: A/H1N1: number analyzed (Participants) | 388 | 386
  Baseline: A/H1N1 | 19.8 [16.0 to 24.2] | 23.6 [19.4 to 28.1]
  4 weeks after vaccination: A/H1N1: number analyzed (Participants) | 390 | 389
  4 weeks after vaccination: A/H1N1 | 70.0 [65.2 to 74.5] | 76.6 [72.1 to 80.7]
  Baseline: B/Yamagata: number analyzed (Participants) | 386 | 385
  Baseline: B/Yamagata | 56.5 [51.4 to 61.5] | 61.0 [56.0 to 65.9]
  4 weeks after vaccination: B/Yamagata: number analyzed (Participants) | 387 | 389
  4 weeks after vaccination: B/Yamagata | 82.9 [78.8 to 86.6] | 87.4 [83.7 to 90.5]
  Baseline: B/Victoria: number analyzed (Participants) | 385 | 382
  Baseline: B/Victoria | 54.8 [49.7 to 59.9] | 50.8 [45.7 to 55.9]
  4 weeks after vaccination: B/Victoria: number analyzed (Participants) | 386 | 382
  4 weeks after vaccination: B/Victoria | 80.8 [76.5 to 84.6] | 86.9 [83.1 to 90.1]

51. Secondary Outcome: HAI GMTs at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: HAI GMTs at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Titers
  Baseline: A/H3N2: number analyzed (Participants) | 382 | 381
  Baseline: A/H3N2 | 32.9 [29.7 to 36.5] | 30.4 [27.4 to 33.7]
  4 Weeks after vaccination: A/H3N2: number analyzed (Participants) | 382 | 381
  4 Weeks after vaccination: A/H3N2 | 224.0 [199.2 to 252.0] | 96.8 [86.2 to 108.7]
  Baseline: A/H1N1: number analyzed (Participants) | 390 | 390
  Baseline: A/H1N1 | 14.8 [13.1 to 16.7] | 15.0 [13.3 to 17.0]
  4 Weeks after vaccination: A/H1N1: number analyzed (Participants) | 390 | 390
  4 Weeks after vaccination: A/H1N1 | 129.5 [111.9 to 149.9] | 88.0 [76.3 to 101.3]
  Baseline: B/Yamagata: number analyzed (Participants) | 389 | 386
  Baseline: B/Yamagata | 16.1 [14.7 to 17.6] | 16.1 [14.7 to 17.6]
  4 Weeks after vaccination: B/Yamagata: number analyzed (Participants) | 389 | 386
  4 Weeks after vaccination: B/Yamagata | 40.4 [37.2 to 43.7] | 38.0 [34.6 to 41.9]
  Baseline: B/Victoria: number analyzed (Participants) | 388 | 390
  Baseline: B/Victoria | 20.4 [18.3 to 22.9] | 19.6 [17.5 to 22.0]
  4 Weeks after vaccination: B/Victoria: number analyzed (Participants) | 388 | 390
  4 Weeks after vaccination: B/Victoria | 45.9 [41.3 to 51.1] | 55.6 [49.6 to 62.4]

53. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for 2023 Southern Hemisphere- Based on HAI Assay 1: 18-64 Years
Time Frame: Before Vaccination (baseline) to 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: HAI GMFR Before Vaccination to 4 Weeks After Vaccination for the 2023 Southern Hemisphere - Based on HAI Assay 1: >=65 Years
Description: GMFRs were defined as ratios of the results after vaccination to the results before vaccination (baseline).
Time Frame: Before vaccination (baseline) to 4 weeks after vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Fold rise
  A/H3N2: number analyzed (Participants) | 382 | 381
  A/H3N2 | 6.4 [5.8 to 7.1] | 3.0 [2.7 to 3.3]
  A/H1N1: number analyzed (Participants) | 390 | 390
  A/H1N1 | 6.8 [6.0 to 7.6] | 4.5 [4.0 to 5.1]
  B/Yamagata: number analyzed (Participants) | 389 | 386
  B/Yamagata | 2.2 [2.1 to 2.3] | 2.1 [1.9 to 2.3]
  B/Victoria: number analyzed (Participants) | 388 | 390
  B/Victoria | 2.0 [1.8 to 2.1] | 2.5 [2.3 to 2.7]

55. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion at 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: 18-64 Years
Time Frame: 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion at 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: >=65 Years
Description: as for outcome 48
Time Frame: 4 weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Percentage of participants
  A/H3N2: number analyzed (Participants) | 382 | 381
  A/H3N2 | 81.7 [77.4 to 85.4] | 44.9 [39.8 to 50.0]
  A/H1N1: number analyzed (Participants) | 390 | 390
  A/H1N1 | 77.2 [72.7 to 81.3] | 57.9 [52.9 to 62.9]
  B/Yamagata: number analyzed (Participants) | 389 | 386
  B/Yamagata | 29.8 [25.3 to 34.6] | 28.8 [24.3 to 33.6]
  B/Victoria: number analyzed (Participants) | 388 | 390
  B/Victoria | 23.5 [19.3 to 28.0] | 36.9 [32.1 to 41.9]

57. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: 18-64 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 43
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 at Baseline and 4 Weeks After Vaccination for 2023 Southern Hemisphere - Based on HAI Assay 1: >=65 Years
Time Frame: Baseline and 4 weeks after vaccination
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | qIRV: >=65 Years | Licensed QIV: >=65 Years
Number analyzed (Participants) | 391 | 390
Percentage of participants
  Baseline: A/H3N2: number analyzed (Participants) | 382 | 381
  Baseline: A/H3N2 | 61.3 [56.2 to 66.2] | 58.3 [53.1 to 63.3]
  4 weeks after vaccination: A/H3N2: number analyzed (Participants) | 382 | 381
  4 weeks after vaccination: A/H3N2 | 98.2 [96.3 to 99.3] | 89.8 [86.3 to 92.6]
  Baseline: A/H1N1: number analyzed (Participants) | 390 | 390
  Baseline: A/H1N1 | 27.9 [23.5 to 32.7] | 28.5 [24.0 to 33.2]
  4 weeks after vaccination: A/H1N1: number analyzed (Participants) | 390 | 390
  4 weeks after vaccination: A/H1N1 | 85.6 [81.8 to 89.0] | 77.9 [73.5 to 82.0]
  Baseline: B/Yamagata: number analyzed (Participants) | 389 | 386
  Baseline: B/Yamagata | 28.5 [24.1 to 33.3] | 26.7 [22.3 to 31.4]
  4 weeks after vaccination: B/Yamagata: number analyzed (Participants) | 389 | 386
  4 weeks after vaccination: B/Yamagata | 69.4 [64.6 to 74.0] | 61.9 [56.9 to 66.8]
  Baseline: B/Victoria: number analyzed (Participants) | 388 | 390
  Baseline: B/Victoria | 38.1 [33.3 to 43.2] | 34.6 [29.9 to 39.6]
  4 weeks after vaccination: B/Victoria: number analyzed (Participants) | 388 | 390
  4 weeks after vaccination: B/Victoria | 69.3 [64.5 to 73.9] | 73.8 [69.2 to 78.1]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events (Systematic assessment): from Day 1 to Day 7 after vaccination; Non-systematic assessment: SAEs: from vaccination 1 up to 6 months after last vaccination, other AEs: from vaccination 1 up to 4 weeks after last vaccination and All-cause mortality: From vaccination on Day 1 up to 6 months after vaccination.
Description: Same adverse event (preferred term) may appear as both non-SAE and SAE but are distinct events. An adverse event (preferred term) may be categorized as serious in 1 participant and non-serious in another. Safety population included all participants who received the study intervention at the specified dose level. Participants were included in the vaccination group corresponding to the study intervention that they actually received.
Groups:
- Licensed QIV: >=18 Years: Participants aged >=18 years were randomized to receive a single dose of seasonal licensed QIV IM per IPM on Day 1.
Arm/Group | qIRV: 18-64 Years | Licensed QIV: 18-64 Years | qIRV: >=65 Years | Licensed QIV: >=65 Years | qIRV (>=18 Years) | Licensed QIV: >=18 Years
All-Cause Mortality (participants affected / at risk) | 7/9191 | 9/9197 | 49/13557 | 46/13611 | 56/22787 | 55/22808
Serious Adverse Events (participants affected / at risk) | 83/9191 | 93/9197 | 318/13557 | 296/13611 | 401/22787 | 389/22808
Other Adverse Events (participants affected / at risk) | 2607/9191 | 1964/9197 | 3091/13557 | 1720/13611 | 5698/22787 | 3684/22808
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | qIRV: 18-64 Years (N=9191) | Licensed QIV: 18-64 Years (N=9197) | qIRV: >=65 Years (N=13557) | Licensed QIV: >=65 Years (N=13611) | qIRV (>=18 Years) (N=22787) | Licensed QIV: >=18 Years (N=22808)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1 | 4 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 3 | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 6 | 10 | 7 | 12
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 0 | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 21 | 15 | 23 | 16
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 3 | 1 | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 2 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2 | 8 | 3 | 8 | 5
Cardiac failure (Cardiac disorders) | 1 | 1 | 3 | 2 | 4 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 3 | 1 | 3 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 2 | 10 | 13 | 12 | 15
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 4 | 5 | 4 | 6
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 9 | 7 | 9 | 7
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 3 | 2 | 3 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 3 | 8 | 7 | 8 | 10
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 2 | 1 | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 3 | 0 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 3 | 0 | 4 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Middle ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 2 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 3 | 5
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Retroperitoneal effusion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 4 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 9 | 1 | 9 | 2
Death (General disorders) | 2 | 0 | 6 | 3 | 8 | 3
Multi-organ disorder (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 4 | 1 | 4 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Organ failure (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 2 | 1 | 4 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 3 | 5 | 3 | 5
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 2 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 2 | 0 | 3 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Amoebic dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 4 | 2 | 2 | 1 | 6 | 3
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 4 | 2 | 4 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 3 | 0 | 3 | 1
Cellulitis (Infections and infestations) | 1 | 3 | 5 | 6 | 6 | 9
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 2 | 4 | 2 | 6 | 4
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 2 | 3 | 2
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 3 | 0 | 3 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Haemophilus bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Infective tenosynovitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 1
Kidney infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 3 | 0 | 3 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 7 | 25 | 25 | 32 | 32
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 3 | 0 | 3 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 2 | 9 | 8 | 11 | 10
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 6 | 7 | 6 | 7
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Submandibular abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 7 | 2 | 7 | 2
Urosepsis (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 5 | 2 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 3 | 4 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 3 | 5 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 2 | 2
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 2 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 1 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 2 | 1
Vaginal cuff dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Human rhinovirus test positive (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 6 | 1 | 6 | 1
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 4 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 2 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 1 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 6 | 4 | 7 | 5
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 1 | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 1 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 2 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 1 | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 2 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 2 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Mueller's mixed tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 2 | 1
Neuroendocrine carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Ocular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 0 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4 | 5 | 6 | 5
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Axonal and demyelinating polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 8 | 9 | 9 | 9
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 3 | 1 | 3
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 3
Idiopathic intracranial hypertension (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 4 | 4 | 4 | 4
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 2 | 2 | 2 | 2
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Myelin oligodendrocyte glycoprotein antibody-associated disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 2 | 2 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Seizure (Nervous system disorders) | 2 | 1 | 3 | 0 | 5 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 2 | 3 | 2 | 4
Syncope (Nervous system disorders) | 0 | 3 | 4 | 3 | 4 | 6
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 6 | 5 | 7 | 5
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 0 | 0 | 2 | 2
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 1 | 0
Device inappropriate shock delivery (Product Issues) | 0 | 0 | 0 | 1 | 0 | 1
Device issue (Product Issues) | 0 | 0 | 0 | 1 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 1 | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 2 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 1 | 1 | 2 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 2 | 0 | 1 | 2 | 3
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dysphemia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 2 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 16 | 7 | 17 | 8
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 4 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 2 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 3 | 3 | 3 | 3
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Renal tubular injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 4 | 2 | 4 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 17 | 6 | 18 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2 | 3 | 3
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 10 | 12 | 12 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2 | 3 | 3
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 4 | 4 | 5
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 5 | 7 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 3 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4 | 1 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Substance use (Social circumstances) | 1 | 0 | 0 | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 2
Aortic dilatation (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2
Aortic embolus (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Aortic intramural haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cyanosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 2 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 2 | 1 | 2
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 2 | 2 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Internal haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Necrosis ischaemic (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Penetrating atherosclerotic ulcer (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 2 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Scalp haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | qIRV: 18-64 Years (N=9191) | Licensed QIV: 18-64 Years (N=9197) | qIRV: >=65 Years (N=13557) | Licensed QIV: >=65 Years (N=13611) | qIRV (>=18 Years) (N=22787) | Licensed QIV: >=18 Years (N=22808)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 355 | 332 | 272 | 237 | 627 | 569
Chills (CHILLS) (General disorders) | 731 | 249 | 580 | 133 | 1311 | 382
Fatigue (FATIGUE) (General disorders) | 1579 | 1046 | 1624 | 812 | 3203 | 1858
Injection site erythema (REDNESS) (General disorders) | 230 | 105 | 376 | 95 | 606 | 200
Injection site pain (General disorders) | 142 | 66 | 274 | 74 | 416 | 140
Injection site pain (PAIN) (General disorders) | 2112 | 1284 | 2391 | 840 | 4503 | 2124
Injection site swelling (SWELLING) (General disorders) | 254 | 129 | 383 | 129 | 637 | 258
Pyrexia (FEVER) (General disorders) | 170 | 52 | 201 | 36 | 371 | 88
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 493 | 208 | 407 | 201 | 900 | 409
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 920 | 307 | 715 | 251 | 1635 | 558
Headache (HEADACHE) (Nervous system disorders) | 1273 | 853 | 1043 | 543 | 2316 | 1396

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT05540522/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT05540522/SAP_001.pdf